CLINICAL TRIAL: NCT07001579
Title: Prevalence and Associated Risk Factors of Asymptomatic Bacteriuria in Pregnancy at a Tertiary Care Hospital: a Cross-sectional Duty
Brief Title: Cross-sectional Study of the Prevalence and Risk Factors of Asymptomatic Bacteriuria in Pregnancy
Status: Completed | Type: Observational
Sponsor: Nepalese Army Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sabin Poudel, Dr., Nepalese Army Institute of Health Sciences
Other Study IDs: SBH-AUTI-2022-01
Record Dates: First submitted 2025-05-07; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Urinary Tract Infection (Diagnosis); Pregnancy
MeSH Terms: conditions — Urinary Tract Infections; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asymptomatic bacteriuria (ASB) is the presence of bacteria in the urine without symptoms of urinary tract infection. It is common during pregnancy and, if left untreated, may lead to complications such as pyelonephritis, preterm labor, and low birth weight. This cross-sectional study aims to determine the prevalence and identify associated risk factors of ASB among pregnant women attending antenatal care at a tertiary care hospital. Pregnant women meeting the inclusion criteria will be enrolled and evaluated through urine analysis and relevant history-taking. The findings may help guide future screening and treatment policies in antenatal care settings

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending her regular ANC check-ups at the hospital.
* Who give consent to participate in the study.

Exclusion Criteria:

* Individuals not willing to participate
* Pregnant women showing signs and symptoms of UTI.
* Pregnant women on antibiotics or had been on antibiotics at least two weeks prior to presentation.
* Pregnant women with known underlying renal pathology.
* Pregnant women who are using immune-suppressants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since, it is study of Asymptomatic Urinary Tract Infection in pregnancy. This involves only female.
Study Population: Pregnant women visiting the Department of Obstetrics and Gynecology OPD, (Shree Birendra Hospital) located in Kathmandu for Antenatal Check-up.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of Asymptomatic Bacteriuria in Pregnant Women | Data was collected for 6 months after approval from IRC from April 2022 to September 2022 during each participant's first antenatal care (ANC) visit irrespective of the gestational age, using simple convenient sampling method.
  The proportion of pregnant women attending antenatal care who test positive for asymptomatic bacteriuria based on urine culture

CONTACTS AND LOCATIONS:
Locations (1):
- Shree Birendra Hospita, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No